CLINICAL TRIAL: NCT01451645
Title: Efficacy and Safety of Colchicine for the Prevention of Gout Flares During the Initiation of Allopurinol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IL1T-GA-1103
Record Dates: First submitted 2011-10-10; First posted 2011-10-14 (Estimated); Results first posted 2014-05-12 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-04

CONDITIONS: Intercritical Gout
Keywords: Gout
MeSH Terms: conditions — Gout | interventions — Colchicine; Allopurinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Other): daily placebo dosing for 16 weeks with background allopurinol therapy
  Interventions: Drug: placebo; Drug: allopurinol
- Colchicine (Colcrys®) (Active Comparator): daily 0.6 mg colchicine dosing for 16 weeks with background allopurinol therapy
  Interventions: Drug: Colchicine (Colcrys®); Drug: allopurinol

INTERVENTIONS:
Drug: Colchicine (Colcrys®) — daily 0.6 mg colchicine dosing for 16 weeks
  Arms: Colchicine (Colcrys®)
Drug: placebo — daily placebo dosing for 16 weeks
  Arms: placebo
Drug: allopurinol — background therapy

SUMMARY:
The purpose of this study is to determine if once-daily treatment with colchicine, compared to placebo, is effective in preventing gout flares in patients who are initiating therapy with allopurinol.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria include, but are not limited to the following:

1. Men and postmenopausal women between the ages of 18 and 70
2. Meets the ARA criteria for classification of acute gout
3. Tophi present and/or a history of gout attacks in 2 or 3 joints
4. Self-reported history of at least 2 gout flares in the prior 12 months
5. Serum uric acid greater than or equal to 7.5 mg/dL at the first visit

Exclusion Criteria:

Exclusion criteria include, but are not limited to the following:

1. Patients with an acute gout flare within 2 weeks prior to the first visit
2. Patients with chronic, active gout with at least 1 continuously inflamed joint for at least 4 weeks
3. Patients with more than three joints affected by gout
4. History of intolerance or allergy to colchicine or allopurinol
5. Use of allopurinol, benzbromarone, febuxostat, probenecid, or sulfinpyrazone less than 3 months prior to entering the study
6. Use of colchicine less than 14 days prior to entering the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2011-10; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (37):
- United States (37):
  - Alabaster, Alabama
  - Mesa, Arizona
  - Upland, California
  - Trumbull, Connecticut
  - DeBary, Florida
  - Jacksonville, Florida
  - Kissimmee, Florida
  - Canton, Georgia
  - Boise, Idaho
  - Lexington, Kentucky
  - Bethesda, Maryland
  - Reisterstown, Maryland
  - Bingham Farms, Michigan
  - Brooklyn Center, Minnesota
  - Kansas City, Missouri
  - Billings, Montana
  - Elizabeth, New Jersey
  - Albuquerque, New Mexico
  - New York, New York
  - Charlotte, North Carolina
  - Hickory, North Carolina
  - Morganton, North Carolina
  - Winston-Salem, North Carolina
  - Duncansville, Pennsylvania
  - Reading, Pennsylvania
  - West Reading, Pennsylvania
  - Greer, South Carolina
  - Mt. Pleasant, South Carolina
  - Johnson City, Tennessee
  - Dallas, Texas
  - Katy, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Norfolk, Virginia
  - Seattle, Washington
  - Wauwatosa, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 82 patients from 20 clinical sites participated in the study between 19-October-2011 to 27-August-2012.
Pre-assignment Details: Participants were assessed at an initial screening visit within 3 to 14 days before the baseline visit. At the baseline visit, eligible participants were then assessed, randomized, trained on daily dosing & the daily dosing/flare diary, and initiated on allopurinol and study drug (colchicine or placebo).
Groups:
- Colchicine (Colcrys®) 0.6mg: daily 0.6 mg colchicine dosing for 16 weeks with background allopurinol therapy
Period: Overall Study
Arm/Group | Placebo | Colchicine (Colcrys®) 0.6mg
Started | 41 | 41
Completed | 32 | 33
Not Completed | 9 | 8
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 0 | 3
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Lost to Follow-up | 4 | 3

BASELINE CHARACTERISTICS:
Population: The study population consisted of adults who met the criteria of the ARA for acute arthritis of primary gout or had monosodium urate monohydrate microcrystals identified in joint fluid, had tophi present in joints or a history of polyarticular gout attacks, a history of ≥2 gout flares in the past year, and were initiating therapy with allopurinol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Colchicine (Colcrys®) 0.6mg | Total
Number analyzed (Participants) | 41 | 41 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 35 | 74
  >=65 years | 2 | 6 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 7
  Male | 40 | 35 | 75

OUTCOME MEASURES:

1. Primary Outcome: Number of Gout Flares Per Participant From Day 1 to Week 16
Time Frame: Day 1 to Week 16
Population: Efficacy endpoints were analyzed using the FAS. The full analysis set (FAS) included all randomized patients who received any study drug; it is based on the treatment allocated (as randomized).
Measure: Mean (Standard Deviation); unit: gout flares
Arm/Group | Placebo | Colchicine (Colcrys®) 0.6mg
Number analyzed (Participants) | 41 | 41
gout flares | 1.1 (1.90) | 0.3 (0.56)

2. Secondary Outcome: Percentage of Participants With at Least 1 Gout Flare From Day 1 to Week 16
Time Frame: Day 1 to Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Colchicine (Colcrys®) 0.6mg
Number analyzed (Participants) | 41 | 41
Percentage of Participants | 43.9 [28.47 to 60.25] | 24.4 [12.36 to 40.30]

3. Secondary Outcome: Percentage of Participants With at Least 2 Gout Flares From Day 1 to Week 16
Time Frame: Day 1 to Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Colchicine (Colcrys®) 0.6mg
Number analyzed (Participants) | 41 | 41
Percentage of Participants | 24.4 [12.36 to 40.30] | 4.9 [0.60 to 16.53]

4. Secondary Outcome: Mean Number of Gout Flare Days Per Participant Assessed From Day 1 to Week 16
Time Frame: Day 1 to Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Colchicine (Colcrys®) 0.6mg
Number analyzed (Participants) | 41 | 41
days | 6.6 (13.20) | 1.6 (3.75)

ADVERSE EVENTS:
Arm/Group | Placebo | Colchicine (Colcrys®) 0.6mg
Serious Adverse Events (participants affected / at risk) | 0/41 | 1/41
Other Adverse Events (participants affected / at risk) | 20/41 | 20/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | Colchicine (Colcrys®) 0.6mg (N=41)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | Colchicine (Colcrys®) 0.6mg (N=41)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Headache (Nervous system disorders) | 7 | 7
Hypoaesthesia (Nervous system disorders) | 0 | 3
Nasopharyngitis (Infections and infestations) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Insomnia (Psychiatric disorders) | 3 | 0

LIMITATIONS AND CAVEATS:
This clinical trial was not directly related to the development of an investigational/medicinal product.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Not less than 45 days prior to submission for publication or presentation, the Institution shall, or cause the Principal Investigator to, provide the Sponsor with a copy of the Manuscript. The Institution shall consider in good faith any comments from the Sponsor regarding the content, and shall delete Confidential Information upon written request of the Sponsor. At the Sponsor's request, the Institution shall delay publication for an additional 60 days to allow patent applications to be filed.